CLINICAL TRIAL: NCT06546293
Title: The Effect of Core Stabilization Training on Pain, Functional Status, Fatigue, and Quality of Life in Patients with Juvenile Spondyloarthropathy
Brief Title: Core Stabilization Training in Juvenile Spondyloarthropathy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Gokce Leblebici, Principal investigator, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IUC_SpA_core
Record Dates: First submitted 2024-08-06; First posted 2024-08-09 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2024-08

CONDITIONS: Spondylarthritis; Spondylarthropathies; Juvenile Idiopathic Arthritis
MeSH Terms: conditions — Spondylarthritis; Spondylarthropathies; Arthritis, Juvenile

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Core stabilization group (Experimental): lumbo-pelvic/core strength and stability exercises group
  Interventions: Other: core stabilization exercises
- Control group (Active Comparator): the group that will have a daily physical activity program established and monitored for participation through weekly exercise tracking chart
  Interventions: Other: daily physical activity program

INTERVENTIONS:
Other: core stabilization exercises — The program consists of lumbo-pelvic/core strength and stability exercises. The program will be implemented individually under the supervision of a physiotherapist twice a week for 12 weeks.
  Arms: Core stabilization group
Other: daily physical activity program — The program consists of a daily physical activity program established and monitored for participation through weekly exercise tracking chart. The program will be implemented through weekly physiotherapist's control of the exercise tracking chart for 12 weeks.
  Arms: Control group

SUMMARY:
Core stabilization exercises developed by McGill have been shown to be one of the physiotherapy techniques aimed at reducing pain, increasing aerobic capacity, enhancing muscle strength, and thereby improving bone health in children with JIA. However, there is no study that has investigated core stabilization training for different types of JIA. In our study, we aim to compare the effectiveness of core stabilization training and a daily physical activity program in children with spondyloarthropathy, to help identify the most effective strategy for clinical practice. Additionally, highlighting the specific effects of core stabilization training on the treatment of juvenile spondyloarthropathy (pain, functional status, fatigue, and quality of life) will make a significant contribution to the literature.

Taking into account the gaps in the literature, our study will investigate the effect of core stabilization training on pain, functional status, fatigue, and quality of life in patients with juvenile spondyloarthropathy.

DETAILED DESCRIPTION:
Core stabilization exercises are one of the physiotherapy techniques aimed at reducing pain, increasing aerobic capacity, enhancing muscle strength, and thereby improving bone health in children with JIA (1). Spondyloarthropathy typically begins as asymmetric oligoarthritis in children, and enthesitis and axial skeleton involvement may develop over the course of the disease (4). Since juvenile spondyloarthropathies can lead to severe functional impairments and long-term sequelae, the primary goal in treatment should be to suppress inflammation as early as possible and to prevent sequelae (5). Physiotherapy is recommended for children and adolescents with enthesitis or sacroiliitis, or those with functional limitations (6). Yoga exercises focusing on the core region have shown significant effects on lower extremity functional status, pain levels, and quality of life in patients with enthesitis-related conditions (2). Studies have supported that core stabilization exercises, combined with traditional physical therapy aimed at improving bone health status and functional capacity, serve as an effective combination therapy for children with JIA involving multiple joint involvement (3).

Therefore, this study aims to fill the knowledge gap regarding core stabilization training in children with spondyloarthropathy.

ELIGIBILITY:
Inclusion Criteria:

* "According to the International League of Associations for Rheumatology criteria, individuals aged 10-18 diagnosed with spondyloarthritis within the JIA subgroup will be included.
* Only cases with stable disease activity and without additional neurological or orthopedic conditions will be considered.
* Participants must also possess the cognitive ability to engage in active rehabilitation.

Exclusion Criteria:

* Individuals with a cardiovascular disease that impedes exercise
* those who have participated in a rehabilitation program within the last 6 months
* cases with variable medical treatment will be excluded.

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale | immediately after intervention
  Pain intensity assessment in the lower extremity regions of the sacroiliac joint, hip, knee, and ankle. It is frequently used to quantify the severity or frequency of different symptoms in epidemiologic and clinical research. From the standpoint of the patient, pain seems to be a continuous spectrum rather than discretely varying, as categories like none, mild, moderate, and severe would imply. To represent this concept of an underlying continuum, the VAS was developed.

SECONDARY OUTCOMES:
Six minute walk test | immediately after intervention
  The general functional status of the lower extremities will be evaluated by measuring the six-minute walking distance. The assessment will be conducted along a 15-meter monitored corridor, and the children will be asked to walk as quickly as possible without running. Standard encouragement instructions such as 'keep going' or 'you are doing well' will be used. The children will be allowed to stop and rest during the test, but the countdown will not be paused in these instances. The distance covered over six minutes will be recorded.
Pediatric quality of life | immediately after intervention
  To assess quality of life, the Turkish version of the Pediatric Quality of Life Inventory (PedsQL) 3.0 Arthritis (Rheumatology) Module will be used. The PedsQL 3.0 Arthritis Module includes a total of 22 questions across five different domains: pain and hurt (4 items), daily activities (5 items), treatment (7 items), worry (3 items), and communication (3 items). The questionnaire is available in two forms: a patient form and a parent form. Both the children and one of their parents will complete the PedsQL 3.0 Arthritis Module.
PedsQL-Multidimensional Fatigue Scale | immediately after intervention
  General fatigue, sleep/rest fatigue, cognitive fatigue, and overall fatigue scores will be assessed. Scoring for all child, adolescent, young adult, and parent surveys is conducted on a five-point Likert scale (0 = Never; 1 = Almost Never; 2 = Sometimes; 3 = Often; 4 = Almost Always). A score of 0 indicates high fatigue, while a score of 100 indicates less fatigue on the PedsQL-MFS item scoring.
Timed Up and Down Stairs Test (TUDS) | immediately after intervention
  The individual taking part is standing one foot from the bottom of a 14-step staircase. "Quickly, but safely, go up the stairs, turn around on the top step (landing), and come all the way down until both feet land on the bottom step," is the participant's instruction.
  The amount of time, measured in seconds, between the "go" signal and the second foot returning to the bottom landing was the TUDS score. Faster times correlated with higher functional proficiency.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University-Cerrahpasa, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] McGill SM, Childs A, Liebenson C. Endurance times for low back stabilization exercises: clinical targets for testing and training from a normal database. Arch Phys Med Rehabil. 1999 Aug;80(8):941-4. doi: 10.1016/s0003-9993(99)90087-4. PMID 10453772
- [Background] Yasar E, Kavlak E, Turkucar S, Bayraktar D, Acari C, Unsal E. Yoga versus home exercise program in children with enthesitis related arthritis: A pilot study. Complement Ther Med. 2021 May;58:102696. doi: 10.1016/j.ctim.2021.102696. Epub 2021 Feb 23. PMID 33636297
- [Background] Elnaggar RK, Mahmoud WS, Moawd SA, Azab AR. Impact of core stability exercises on bone mineralization and functional capacity in children with polyarticular juvenile idiopathic arthritis: a randomized clinical trial. Clin Rheumatol. 2021 Jan;40(1):245-253. doi: 10.1007/s10067-020-05219-9. Epub 2020 Jun 8. PMID 32514677
- [Background] Weiss PF, Roth J. Juvenile-Versus Adult-Onset Spondyloarthritis: Similar, but Different. Rheum Dis Clin North Am. 2020 May;46(2):241-257. doi: 10.1016/j.rdc.2020.01.003. PMID 32340699
- [Background] Yildiz M, Haslak F, Adrovic A, Sahin S, Barut K, Kasapcopur O. Juvenile spondyloartropathies. Eur J Rheumatol. 2022 Jan;9(1):42-49. doi: 10.5152/eurjrheum.2021.20235. PMID 34101576
- [Background] Ringold S, Angeles-Han ST, Beukelman T, Lovell D, Cuello CA, Becker ML, Colbert RA, Feldman BM, Ferguson PJ, Gewanter H, Guzman J, Horonjeff J, Nigrovic PA, Ombrello MJ, Passo MH, Stoll ML, Rabinovich CE, Schneider R, Halyabar O, Hays K, Shah AA, Sullivan N, Szymanski AM, Turgunbaev M, Turner A, Reston J. 2019 American College of Rheumatology/Arthritis Foundation Guideline for the Treatment of Juvenile Idiopathic Arthritis: Therapeutic Approaches for Non-Systemic Polyarthritis, Sacroiliitis, and Enthesitis. Arthritis Rheumatol. 2019 Jun;71(6):846-863. doi: 10.1002/art.40884. Epub 2019 Apr 25. PMID 31021537
- [Background] Miro J, Castarlenas E, de la Vega R, Sole E, Tome-Pires C, Jensen MP, Engel JM, Racine M. Validity of three rating scales for measuring pain intensity in youths with physical disabilities. Eur J Pain. 2016 Jan;20(1):130-7. doi: 10.1002/ejp.704. Epub 2015 Mar 31. PMID 25833415
- [Background] Lelieveld OT, Takken T, van der Net J, van Weert E. Validity of the 6-minute walking test in juvenile idiopathic arthritis. Arthritis Rheum. 2005 Apr 15;53(2):304-7. doi: 10.1002/art.21086. No abstract available. PMID 15818658
- [Background] Zaino CA, Marchese VG, Westcott SL. Timed up and down stairs test: preliminary reliability and validity of a new measure of functional mobility. Pediatr Phys Ther. 2004 Summer;16(2):90-8. doi: 10.1097/01.PEP.0000127564.08922.6A. PMID 17057533
- [Background] Tarakci E, Baydogan SN, Kasapcopur O, Dirican A. Cross-cultural adaptation, reliability, and validity of the Turkish version of PedsQL 3.0 Arthritis Module: a quality-of-life measure for patients with juvenile idiopathic arthritis in Turkey. Qual Life Res. 2013 Apr;22(3):531-6. doi: 10.1007/s11136-012-0180-0. Epub 2012 Apr 29. PMID 22544413